CLINICAL TRIAL: NCT00184795
Title: A Six Month Double-blind, Randomised, Parallel-group, Placebo-controlled, Multi-centre Trial to Investigate the Efficacy and Safety of Two Ultra-low Dose Combinations With 0.5 mg Estradiol and 0.1 mg or 0.25 mg Norethisterone Acetate (Activelle Low Dose 0.1/Activelle Low Dose 0.25) for Treatment of Menopausal Symptoms
Brief Title: Bleed Free Treatment of Menopausal Symptoms With New Ultra Low Dose Hormonal Combinations
Acronym: CHOICE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALD-1537; 2004-000103-17 (EudraCT Number)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Menopause; Menopausal Vasomotor Symptoms
Keywords: Hot flashes
MeSH Terms: conditions — Hot Flashes | interventions — Estradiol; Norethindrone Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ALD 0.1 (Experimental)
  Interventions: Drug: 0.5 mg estradiol / 0.1 mg norethisterone acetate (NETA)
- ALD 0.25 (Experimental)
  Interventions: Drug: 0.5 mg estradiol / 0.25 mg norethisterone acetate (NETA)
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 0.5 mg estradiol / 0.1 mg norethisterone acetate (NETA) — One tablet per day for 24 weeks
  Arms: ALD 0.1
Drug: 0.5 mg estradiol / 0.25 mg norethisterone acetate (NETA) — One tablet per day for 24 weeks
  Arms: ALD 0.25
Drug: placebo — Placebo tablets for 24 weeks
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. Postmenopausal women with moderate to severe hot flashes have been recruited into the trial. The earliest effect of ultra low dose HRT (hormone replacement therapy) on frequency and severity of menopausal symptoms, bleeding patterns and safety of different hormonal combinations will be evaluated and compared to placebo over the six month treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal status
* Subject should have had a minimum of 7 moderate to severe hot flushes per day, or a minimum of 50 moderate to severe hot flushes per week, during the last 2 weeks of the run-in (screening) period.
* Subject with an intact uterus

Exclusion Criteria:

* In accordance with existing labelling for estrogen/progestogen combinations
* Body Mass Index (BMI) > 35.0 kg/m2
* Known alcohol or drug abuse, heavy smoking (more than 20 cigarettes a day)
* Currently using steroid hormones (except topical or inhalation glucocorticoid preparations) and drugs known to influence estrogen metabolism such as barbiturates, phenytoin, rifampicin, carbamazepin

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2004-05-28 (Actual); Primary Completion 2005-05-04 (Actual); Study Completion 2005-05-04 (Actual)

PRIMARY OUTCOMES:
Change in mean number of moderate to severe hot flushes per week | At week 8

SECONDARY OUTCOMES:
Urogenital symptoms | Week 0; week 24
Vaginal cytology and pH | Week 0; week 24
Bleeding profile | Week 0; week 24
Adverse Events | Week 0; week 24
Menopausal symptoms and quality of life (Greene Climacteric Scale) | Week 0; week 24
Hot flush weekly weighted score | Week 0; week 24

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (80):
- Novo Nordisk Investigational Site, Vienna, Austria
- Belgium (7):
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Ghent
  - Novo Nordisk Investigational Site, Huy
  - Novo Nordisk Investigational Site, Leuven
  - Novo Nordisk Investigational Site, Liège
  - Novo Nordisk Investigational Site, Montigny-le-Tilleul
  - Novo Nordisk Investigational Site, Watermael-Boifort
- Denmark (8):
  - Novo Nordisk Investigational Site, Allerød Municipality
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Frederiksberg
  - Novo Nordisk Investigational Site, Hvidovre
  - Novo Nordisk Investigational Site, København N
  - Novo Nordisk Investigational Site, Næstved
  - Novo Nordisk Investigational Site, Odense C
  - Novo Nordisk Investigational Site, Virum
- Finland (5):
  - Novo Nordisk Investigational Site, Espoo
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Tampere
  - Novo Nordisk Investigational Site, Turku
- France (9):
  - Novo Nordisk Investigational Site, Amiens
  - Novo Nordisk Investigational Site, La Roche-sur-Yon
  - Novo Nordisk Investigational Site, Marseille
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Nantes
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nice
  - Novo Nordisk Investigational Site, Nîmes
  - Novo Nordisk Investigational Site, Toulouse
- Germany (10):
  - Novo Nordisk Investigational Site, Jessen
  - Novo Nordisk Investigational Site, Karlsruhe
  - Novo Nordisk Investigational Site, Leipzig
  - Novo Nordisk Investigational Site, Lorsch
  - Novo Nordisk Investigational Site, Rheine
  - Novo Nordisk Investigational Site, Rheinstetten
  - Novo Nordisk Investigational Site, Schorndorf
  - Novo Nordisk Investigational Site, Stuttgart
  - Novo Nordisk Investigational Site, Tübingen
  - Novo Nordisk Investigational Site, Völklingen
- Norway (8):
  - Novo Nordisk Investigational Site, Grålum
  - Novo Nordisk Investigational Site, Hamar
  - Novo Nordisk Investigational Site, Kolbotn
  - Novo Nordisk Investigational Site, Lillestrøm
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Paradis
  - Novo Nordisk Investigational Site, Stavanger
  - Novo Nordisk Investigational Site, Trondheim
- Sweden (6):
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Linköping
  - Novo Nordisk Investigational Site, Lund
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Norrköping
  - Novo Nordisk Investigational Site, Uppsala
- Switzerland (4):
  - Novo Nordisk Investigational Site, Bulle
  - Novo Nordisk Investigational Site, Frauenfeld
  - Novo Nordisk Investigational Site, Weinfelden
  - Novo Nordisk Investigational Site, Zurich
- United Kingdom (22):
  - Novo Nordisk Investigational Site, Aldershot
  - Novo Nordisk Investigational Site, Bexhill-on-Sea
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Bolton
  - Novo Nordisk Investigational Site, Chesterfield, Derbyshire
  - Novo Nordisk Investigational Site, Chippenham
  - Novo Nordisk Investigational Site, Cornwell
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Devon
  - Novo Nordisk Investigational Site, Hastings
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Linclolshire
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Norfolk
  - Novo Nordisk Investigational Site, Oxford
  - Novo Nordisk Investigational Site, Reading
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Stoke-on-Trent
  - Novo Nordisk Investigational Site, Suffolk
  - Novo Nordisk Investigational Site, Watford

REFERENCES:
- [Result] Sturdee DW, Archer DF, Rakov V, Lang E; CHOICE Study Investigators. Ultra-low-dose continuous combined estradiol and norethisterone acetate: improved bleeding profile in postmenopausal women. Climacteric. 2008 Feb;11(1):63-73. doi: 10.1080/13697130701852390. PMID 18202966
- [Result] Lundstrom E, Bygdeson M, Svane G, Azavedo E, von Schoultz B. Neutral effect of ultra-low-dose continuous combined estradiol and norethisterone acetate on mammographic breast density. Climacteric. 2007 Jun;10(3):249-56. doi: 10.1080/13697130701385805. PMID 17487652
- [Result] Panay N, Ylikorkala O, Archer DF, Gut R, Lang E. Ultra-low-dose estradiol and norethisterone acetate: effective menopausal symptom relief. Climacteric. 2007 Apr;10(2):120-31. doi: 10.1080/13697130701298107. PMID 17453860
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com